CLINICAL TRIAL: NCT04250454
Title: Protocol of a Two-group Open-label Randomized Clinical Trial With Blinded Assessment for Prevention of Contractures in Infants With High Risk of Cerebral Palsy.
Brief Title: Early Intervention in Infants With Cerebral Palsy
Acronym: CONTRACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Elsass Foundation (Other)
Responsible Party: Principal Investigator, Maria Willerslev-Olsen, Ph.d, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CONTRACT333
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cerebral Palsy
Keywords: Early intervention; Contractures
MeSH Terms: conditions — Cerebral Palsy; Contracture | interventions — Contracts

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Elsass Standard Care
- Intervention (Active Comparator): Enriched eviroment, Feed back training, Electrical stimulation, nutrition
  Interventions: Behavioral: CONTRACT

INTERVENTIONS:
Behavioral: CONTRACT — The intervention will consist of four elements:
  1. Personal meeting - detailed information to the parents before the age of 15 weeks CA (1-3 days)
  2. Home Activity Plan (HAP)
  3. Home-based Feedback training
  4. Electrical muscle stimulation
  Combination of these elements has been chosen in order to ensure that optimal muscle growth is achieved through multi-modal stimulation of the motor and cognitive development of the child.
  Arms: Intervention

SUMMARY:
Contractures are a frequent cause of reduced mobility in children with Cerebral palsy (CP) already at the age of 2-3 years. Reduced muscle use and muscle growth have been suggested as key factors in the development of contractures, suggesting that efficient early prevention will have to involve stimuli that can facilitate muscle growth already before the age of 1 year. The present study protocol was developed to assess the effectiveness of an early intervention program, CONTRACT, on muscle growth and mobility in children at very high risk of CP compared with best standard care.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common cause of motor and cognitive disabilities in childhood affecting around 1 out of 500 newborn infants. Contractures and joint deformities are frequent complications, which limit the functional abilities of the children from an early age and are a main life-long challenge for social integration and participation. The functional limitations imposed by the combination of weak paretic muscles and contractures in early childhood also reduce the child´s possibilities of active exploration of its environment and social interaction with its peers. This may have secondary impact on cognitive development and cognitive performance later in life.

Therefore, early intervention to prevent contractures is pivotal in helping motor and cognitive development in children with CP and thereby enable social integration and optimal cognitive and motor performance throughout their life time. The importance of prevention of contractures is also emphasized by the realization that none of the surgical, medical or physical therapies that we have available provide an efficient treatment of contractures once they have become manifest and interfere with joint mobility.

There is growing evidence that reduced growth of muscles is a key factor in the development of contractures. If muscles fail to grow at the same rate as bones they will be subjected to abnormal tension. This and the lack of muscle use may stimulate growth of connective tissue in the muscles causing a stiffer extracellular matrix. Growth of the medial gastrocnemius muscle in infants with CP deviates from that of typically developing (TD) infants around the age of 12-15 month. Pathologically increased stiffness of the muscle tissue is seen some months later consistent with a causal relation between reduced growth and increased stiffness. These findings indicate that efficient prevention of contractures will have to take place before the age of one years and will need to focus on stimulation of muscle growth as a key factor.

Muscle growth depends crucially on muscle use, which is the exact challenge that infants with CP are faced with. How do we get a child who has difficulty activating its muscles to do so when that child has no prior experience of using its muscles and limbs and has little verbal understanding of what it is we want it to do? There is now evidence to support that the early development of the motor system is highly plastic and depends crucially on activity-dependent interaction with the environment. Experimental evidence from kittens and rodents support the existence of a sensitive period soon after birth where descending connections from the motor cortex to the spinal cord are re-organized in an activity-dependent manner. Functional deficits in mature animals who have received central motor lesions prior to or in relation to birth appear to depend on the extent to which this activity-dependent re-organization takes place during the sensitive period. It is unknown whether a similar sensitive period exists in humans, but there is reason to believe that the first 5-6 month after birth constitute a period where the motor system undergo rapid changes that may resemble the sensitive period in rodents and kittens. This period is characterized in humans by so-called fidgety movements (FM) which may reflect a ´calibration´ of the sensori-motor system, where descending connections are re-organized similar to what is seen in animals. Children also acquire the ability of goal-directed movements using visual feedback during this period, which may be related to maturation of the connections from motor cortex to the spinal cord. There is also evidence that 5-6 month old children have acquired a sense of agency over their own movements and a basic understanding of how they may use their body to control their environment. Sensory feedback and reward that are associated to successful behavior play an important role in this early establishment of movement control. Thelen & Fissher showed that when infants at an very early age can activate a mobile by own spontaneous movements, movement of the infant increased. The initial 5-6 month after term may therefore provide a window of opportunity where it is possible to facilitate normal development of movement and thereby also prevent contractures through the concomitant muscle growth-stimulus. An intervention in which infants in that age group are stimulated to move by their parents at home under supervision by therapists has indeed been demonstrated to improve motor development in infants with high risk of cerebral palsy. Home-training technology that may facilitate the training and the interaction between therapists and the families are also now becoming available and have shown promising effects on motor development in preterm infants . Intensive goal-oriented training involving experiences of success and frequent reward within the first 5-6 month is therefore central in the intervention that we propose in the present protocol for prevention of contractures in infants at high risk of developing CP.

Muscle growth does not only depend on neural and mechanical stimuli, but also on nutritional and metabolic stimuli. It is therefore important also to consider the nutritional status of the infant and especially whether nutrients that have a specific muscle growth promoting effect are delivered in sufficient quantity to the infant either through breast feeding or breast milk substitutes. The polyunsaturated fatty acid, Docosahexaenic acid (DHA) is considered essential for maturation of the developing brain and may also facilitate muscle growth. Supplementation with DHA is not recommended for healthy term-born infants, but may be important for development of preterm infants and especially for infants with brain lesion. In addition, Vitamin D also plays a role in regulating muscle growth and deficiency of Vitamin D has been suggested to be of importance in neurodevelopmental disorders. It is not clear whether early Vitamin D supplementation has beneficial effects on neurodevelopment and muscle growth, but is recommended for newborns in countries with limited sun exposure because of its beneficial effects on bone metabolism. Information about the nutritional status of mother and infant and subsequent supplementation could therefore be of importance to enhance facilitation of muscle growth in the infants.

It should also be considered whether stimuli that may substitute the neural activation of the muscles such as electrical stimulation may be used when the child is not otherwise active (for instance during sleep) to help maintain muscle growth. Electrical muscle stimulation has been shown to diminish muscle atrophy in adults. The facilitation of muscle growth may help to postpone contracture development until communication with the (older) infant is easier and training goals may therefore be achieved more easily.

The purpose of the present paper is consequently to describe a study protocol for a two-group open-label randomized clinical trial with blinded assessment of an early intervention program directed towards prevention of contractures.

ELIGIBILITY:
Inclusion Criteria:

* Infants younger than 17 weeks CA with suspicion of brain lesion determined from a medical assessment, by MRI or ultrasound scan or abcent fidgety movements (FM) determined as part of General Movement Asessement (GMA) will be included. The brain lesion should be rated severe enough by the clinician to have informed the parents of the associated risk of CP.

Exclusion Criteria:

* Infants otherwise eligible but with severe genetic abnormalties, severe heart problems, metabolic diseases, or still hospitalized will not be selected for the study.

Ages: 8 Weeks to 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Muscle growth rate | 48 months
  The primary outcome measure is the rate of muscle growth in the children evaluated from the start of the study until the final end point measurement at 48 month.
  Researchers with high experience in the use of ultrasound (US) examines the entire length of the MG muscle to assess muscle volume. Height, weight, circumference of the widest part of the crus and fibula length is measured. US is performed on the most affected leg or if possible, on both legs, with the infant's ankle fixed in a neutral angle. To estimate muscle thickness and fascicle length one recording is performed with the probe positioned longitudinally at the mid-belly of the MG, with the infant's ankle fixed in a 90-degree angle. The probe was hand-held and fixed vertically with the lower leg for all images.

SECONDARY OUTCOMES:
Evaluation of passive stiffness and reflex stiffness | 48 months
  Passive and reflex-mediated stiffness of the ankle plantar-flexors will be objectively assessed according to the methods described in Lorentzen et al. (Lorentzen et al 2010) and Willerslev-Olsen et al (Willerslev-Olsen et al 2018). Data will be sampled at a rate of 512Hz and transferred to a computer via Bluetooth for further analysis in Matlab (Mathworks, Natick, MA, USA).
  With the use of the device the researcher will move the ankle joint from maximal plantar flexed position to maximal dorsiflexion in order for the devise to estimate the ROM. Manual movements will then be performed by the researcher at either a slow velocity (~<20deg/sec) or as fast as possible through the entire ROM. EMG activity is sampled from bipolar surface EMG electrodes (0.5mm diameter, 2cm between electrodes; Ambu Blue Sensor NF-00-S/12; Ambu, Ballerup, Denmark) placed over the soleus muscle at the distal part of the gastrocnemius muscles and the Tibialis Anterior muscle. The device is equipped with strain

CONTACTS AND LOCATIONS:
Locations (1):
- Elsass Foundation, Charlottenlund, København City, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The university of Copenhagen has a data server available for open acces to research data. We aim to make all annonymised data available through the server as soon as the study has been published in a peer reviewed scientific journal.
Supporting Information: Study Protocol, CSR
Time Frame: When the study has been published in a peer reviewed scientific journal.
Access Criteria: University affiliation

REFERENCES:
- [Background] Rosenbaum P. The natural history of gross motor development in children with cerebral palsy aged 1 to 15 years. Dev Med Child Neurol. 2007 Oct;49(10):724. doi: 10.1111/j.1469-8749.2007.00724.x. No abstract available. PMID 17880638
- [Background] Hagglund G, Wagner P. Spasticity of the gastrosoleus muscle is related to the development of reduced passive dorsiflexion of the ankle in children with cerebral palsy: a registry analysis of 2,796 examinations in 355 children. Acta Orthop. 2011 Dec;82(6):744-8. doi: 10.3109/17453674.2011.618917. Epub 2011 Sep 6. PMID 21895507
- [Background] Shikako-Thomas K, Majnemer A, Law M, Lach L. Determinants of participation in leisure activities in children and youth with cerebral palsy: systematic review. Phys Occup Ther Pediatr. 2008 May;28(2):155-69. doi: 10.1080/01942630802031834. PMID 18846895
- [Background] Spittle A, Orton J, Anderson PJ, Boyd R, Doyle LW. Early developmental intervention programmes provided post hospital discharge to prevent motor and cognitive impairment in preterm infants. Cochrane Database Syst Rev. 2015 Nov 24;2015(11):CD005495. doi: 10.1002/14651858.CD005495.pub4. PMID 26597166
- [Background] Tedroff K, Lowing K, Jacobson DN, Astrom E. Does loss of spasticity matter? A 10-year follow-up after selective dorsal rhizotomy in cerebral palsy. Dev Med Child Neurol. 2011 Aug;53(8):724-9. doi: 10.1111/j.1469-8749.2011.03969.x. Epub 2011 May 18. PMID 21585367
- [Background] Guzzetta A, Mercuri E, Rapisardi G, Ferrari F, Roversi MF, Cowan F, Rutherford M, Paolicelli PB, Einspieler C, Boldrini A, Dubowitz L, Prechtl HF, Cioni G. General movements detect early signs of hemiplegia in term infants with neonatal cerebral infarction. Neuropediatrics. 2003 Apr;34(2):61-6. doi: 10.1055/s-2003-39597. PMID 12776225
- [Background] Willerslev-Olsen M, Choe Lund M, Lorentzen J, Barber L, Kofoed-Hansen M, Nielsen JB. Impaired muscle growth precedes development of increased stiffness of the triceps surae musculotendinous unit in children with cerebral palsy. Dev Med Child Neurol. 2018 Jul;60(7):672-679. doi: 10.1111/dmcn.13729. Epub 2018 Mar 24. PMID 29573407
- [Background] Williams PTJA, Jiang YQ, Martin JH. Motor system plasticity after unilateral injury in the developing brain. Dev Med Child Neurol. 2017 Dec;59(12):1224-1229. doi: 10.1111/dmcn.13581. Epub 2017 Oct 3. PMID 28972274
- [Background] Herskind A, Ritterband-Rosenbaum A, Willerslev-Olsen M, Lorentzen J, Hanson L, Lichtwark G, Nielsen JB. Muscle growth is reduced in 15-month-old children with cerebral palsy. Dev Med Child Neurol. 2016 May;58(5):485-91. doi: 10.1111/dmcn.12950. Epub 2015 Oct 28. PMID 26510820
- [Background] Willerslev-Olsen M, Lorentzen J, Sinkjaer T, Nielsen JB. Passive muscle properties are altered in children with cerebral palsy before the age of 3 years and are difficult to distinguish clinically from spasticity. Dev Med Child Neurol. 2013 Jul;55(7):617-23. doi: 10.1111/dmcn.12124. Epub 2013 Mar 20. PMID 23517272
- [Background] Ritterband-Rosenbaum A, Justiniano MD, Nielsen JB, Christensen MS. Are sensorimotor experiences the key for successful early intervention in infants with congenital brain lesion? Infant Behav Dev. 2019 Feb;54:133-139. doi: 10.1016/j.infbeh.2019.02.001. Epub 2019 Feb 12. PMID 30769300
- [Derived] Willerslev-Olsen M, Lorentzen J, Rohder K, Ritterband-Rosenbaum A, Justiniano M, Guzzetta A, Lando AV, Jensen AB, Greisen G, Ejlersen S, Pedersen LZ, Andersen B, Lipthay Behrend P, Nielsen JB. COpenhagen Neuroplastic TRaining Against Contractures in Toddlers (CONTRACT): protocol of an open-label randomised clinical trial with blinded assessment for prevention of contractures in infants with high risk of cerebral palsy. BMJ Open. 2021 Jul 6;11(7):e044674. doi: 10.1136/bmjopen-2020-044674. PMID 34230015